CLINICAL TRIAL: NCT04648332
Title: Compartment Psoas Block Efficacy and Safety for Perioperative Analgesia in the Elderly With Proximal Femur Fractures: a Randomized Controlled Study
Brief Title: Compartment Psoas Block Efficacy and Safety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bogomolets National Medical University (Other)
Responsible Party: Principal Investigator, Kateryna Bielka, Assistant professor at the Department of OF SURGERY, ANESTHESIOLOGY AND INTENSIVE THERAPY OF POSTGRADUATE EDUCATION, Bogomolets National Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H35LP44qr9
Record Dates: First submitted 2020-09-21; First posted 2020-12-01 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Femur Fracture
Keywords: сompartment psoas block, femur fracture.
MeSH Terms: conditions — Femoral Fractures | interventions — Bupivacaine; Anesthesia, Conduction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): Patients in group 1 underwent catheterization of the lumbar plexus from the posterior access on admission to the hospital and began analgesia with bupivacaine 0.125% 6-8 ml / h. Intraoperative anaesthesia was provided with a bupivacaine bolus of 0.5% 200 mg in a lumbar catheter and a sciatic nerve block with 1.5% 450 mg of lidocaine. Postoperative analgesia was provided by an elongated lumbar plexus block with bupivacaine 0.125% 6-8 ml / h.
  Interventions: Drug: Bupivacaine Hydrochloride
- Group 2 (No Intervention): Patients in group 2 underwent intraoperative spinal anaesthesia at the level of L3-L4 with hyperbaric bupivacaine at a dose of 10-15 mg.
- Group 3 (No Intervention): Group 3 patients underwent general inhalation anaesthesia with sevoflurane with a constant infusion of fentanyl for analgesia.

INTERVENTIONS:
Drug: Bupivacaine Hydrochloride — compartment psoas block
  Other Names: regional anesthesia; compartment psoas block
  Arms: Group 1

SUMMARY:
A randomized controlled trial to assess the efficacy and safety of the prolonged compartment psoas block for analgesia and anesthesia for femur surgery in the elderly

DETAILED DESCRIPTION:
A randomized controlled trial was conducted from January 2018 to August 2019 at the Into-Sana Medical Center (Odessa, Ukraine). The study design was approved by the Ethical Committee at Bogomolets National Medical University. Patients who planned osteosynthesis of the proximal femur and who met the inclusion criteria were randomized to 3 study groupsThe aim of our study was to compare the effectiveness and safety of different techniques of perioperative anaesthesia and anaesthesia in patients with fractures of the proximal femur: general anaesthesia and systemic analgesia, neuraxial (spinal) anaesthesia, compartment psoas block in combination with a sciatic nerve block. Patients in group 1 underwent catheterization of the lumbar plexus from the posterior access on admission to the hospital and began analgesia with bupivacaine 0.125% 6-8 ml / h. Intraoperative anesthesia was provided with a bupivacaine bolus of 0.5% 200 mg in a lumbar catheter and a sciatic nerve block with 1.5% 450 mg of lidocaine. Postoperative analgesia was provided with prolonged lumbar plexus block with bupivacaine 0.125% 6-8 ml / h.

Patients in group 2 underwent intraoperative spinal anaesthesia at the level of L3-L4 with hyperbaric bupivacaine 10-15 mg. Patients in groups 1 - 2 receive intraoperative sedation with propofol 1% with a target level of sedation RASS from 0 to -2. Group 3 patients underwent general sevoflurane inhalation anaesthesia with fentanyl infusion for analgesia.

All patients received paracetamol 3g/day and dexketoprofen 75 mg/day during hospitalization. On-demand, nalbuphine 5 mg SC was used for analgesia.

ELIGIBILITY:
Inclusion Criteria:

-proximal femur fracture

Exclusion Criteria:

* pregnancy and lactation
* history of opiate addiction
* traumatic brain injury
* acute cerebrovascular accident
* chronic heart failure (New York Heart Association Functional Classification, NYHA, class III-IV)
* respiratory failure
* renal failure with decreased creatinine clearance less than 30 ml / min / 1.73 m2
* hepatic insufficiency class C according to Child-Pugh).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
postoperative nalbuphine consumption during first 24 hours and cumulative during hospital stay | 72 hours
  postoperative nalbuphine consumption during first 24 hours and cumulative during hospital stay

SECONDARY OUTCOMES:
ICU length of stay and the total duration of hospitalization | 102 hours
  ICU length of stay and the total duration of hospitalization
number of patients who had severe pain after surgery | 72 hours
  number of patients who had severe pain after surgery
incidence of on-demand analgesia | 72 hours
  incidence of on-demand analgesia

CONTACTS AND LOCATIONS:
Overall Officials: Iurii Kuchyn, PhD, Study Director — Bogomolets National Medical University
Locations (1):
- Bogomolets NMU, Kyiv, Ukraine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cheng SY, Levy AR, Lefaivre KA, Guy P, Kuramoto L, Sobolev B. Geographic trends in incidence of hip fractures: a comprehensive literature review. Osteoporos Int. 2011 Oct;22(10):2575-86. doi: 10.1007/s00198-011-1596-z. Epub 2011 Apr 12. PMID 21484361
- [Background] Dixon J, Ashton F, Baker P, Charlton K, Bates C, Eardley W. Assessment and Early Management of Pain in Hip Fractures: The Impact of Paracetamol. Geriatr Orthop Surg Rehabil. 2018 Oct 25;9:2151459318806443. doi: 10.1177/2151459318806443. eCollection 2018. PMID 30377550
- [Background] Zhang X, Zhou Y, Chen L, Wang Q, Ni J, Liu L, Hu C, Xu X. Anesthesia and postoperative analgesia during unilateral lower-extremity fracture surgeries using multiple injections through catheters beside the lumbar plexus or sciatic nerve. Ther Clin Risk Manag. 2013;9:299-302. doi: 10.2147/TCRM.S45053. Epub 2013 Jul 23. PMID 23901277
- [Background] Demirel I, Ozer AB, Duzgol O, Bayar MK, Karakurt L, Erhan OL. Comparison of unilateral spinal anesthesia and L(1) paravertebral block combined with psoas compartment and sciatic nerve block in patients to undergo partial hip prosthesis. Eur Rev Med Pharmacol Sci. 2014;18(7):1067-72. PMID 24763888
- [Background] Writing Committee for the VISION Study Investigators; Devereaux PJ, Biccard BM, Sigamani A, Xavier D, Chan MTV, Srinathan SK, Walsh M, Abraham V, Pearse R, Wang CY, Sessler DI, Kurz A, Szczeklik W, Berwanger O, Villar JC, Malaga G, Garg AX, Chow CK, Ackland G, Patel A, Borges FK, Belley-Cote EP, Duceppe E, Spence J, Tandon V, Williams C, Sapsford RJ, Polanczyk CA, Tiboni M, Alonso-Coello P, Faruqui A, Heels-Ansdell D, Lamy A, Whitlock R, LeManach Y, Roshanov PS, McGillion M, Kavsak P, McQueen MJ, Thabane L, Rodseth RN, Buse GAL, Bhandari M, Garutti I, Jacka MJ, Schunemann HJ, Cortes OL, Coriat P, Dvirnik N, Botto F, Pettit S, Jaffe AS, Guyatt GH. Association of Postoperative High-Sensitivity Troponin Levels With Myocardial Injury and 30-Day Mortality Among Patients Undergoing Noncardiac Surgery. JAMA. 2017 Apr 25;317(16):1642-1651. doi: 10.1001/jama.2017.4360. PMID 28444280
- [Background] Marufu TC, White SM, Griffiths R, Moonesinghe SR, Moppett IK. Prediction of 30-day mortality after hip fracture surgery by the Nottingham Hip Fracture Score and the Surgical Outcome Risk Tool. Anaesthesia. 2016 May;71(5):515-21. doi: 10.1111/anae.13418. Epub 2016 Mar 4. PMID 26940757
- [Background] White SM, Moppett IK, Griffiths R, Johansen A, Wakeman R, Boulton C, Plant F, Williams A, Pappenheim K, Majeed A, Currie CT, Grocott MP. Secondary analysis of outcomes after 11,085 hip fracture operations from the prospective UK Anaesthesia Sprint Audit of Practice (ASAP-2). Anaesthesia. 2016 May;71(5):506-14. doi: 10.1111/anae.13415. Epub 2016 Mar 4. PMID 26940645
- [Background] Rowlands M, Walt GV, Bradley J, Mannings A, Armstrong S, Bedforth N, Moppett IK, Sahota O. Femoral Nerve Block Intervention in Neck of Femur Fracture (FINOF): a randomised controlled trial. BMJ Open. 2018 Apr 10;8(4):e019650. doi: 10.1136/bmjopen-2017-019650. PMID 29643155
- [Derived] Bielka K, Kuchyn I, Tokar I, Artemenko V, Kashchii U. Psoas compartment block efficacy and safety for perioperative analgesia in the elderly with proximal femur fractures: a randomized controlled study. BMC Anesthesiol. 2021 Oct 25;21(1):252. doi: 10.1186/s12871-021-01473-9. PMID 34696733